CLINICAL TRIAL: NCT01379456
Title: The Effect on Gait and Activity Level of a Physiotherapy Intervention Aimed at Improving Mediolateral Stability 4 Months After a Hip Fracture
Brief Title: Eva-Hip, Evaluation of Rehabilitation After Hip-fracture
Acronym: Eva-Hip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Trondheim Kommune (Other); Norsk kvinners sanitetsforening (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REK 2010/3265-3
Record Dates: First submitted 2011-06-15; First posted 2011-06-23 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physiotherapy (Experimental): exercises
  Interventions: Procedure: physiotherapy
- conventional treatment (No Intervention): care as usual

INTERVENTIONS:
Procedure: physiotherapy — exercises, 20 sessions over 10 weeks
  Arms: physiotherapy

SUMMARY:
To evaluate the effect on gait and activity of a home based physiotherapy intervention 4-6 months after the fracture. The investigators hypothesis is that exercises performed after the initial rehabilitation, which focuses on specific components of gait control will improve gait and increase level of activity.

ELIGIBILITY:
Inclusion Criteria:

* Home dwelling prior to fracture
* age>70yr
* able to walk 10m

Exclusion Criteria:

* expected life expectancies <3 months
* exercises contraindicated due to medical conditions

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 223 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
change in gait speed | 4,6 and 12 months postfracture

SECONDARY OUTCOMES:
change in activity level | 4,6 and 12 month postfracture

CONTACTS AND LOCATIONS:
Overall Officials: Olav Sletvold, MD,PHD, Principal Investigator — Department of Neuroscience, Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Background] Thingstad P, Taraldsen K, Hagen G, Sand S, Saltvedt I, Sletvold O, Helbostad JL. Effectiveness of task specific gait and balance exercise 4 months after hip fracture: protocol of a randomized controlled trial--the Eva-hip study. Physiother Res Int. 2015 Jun;20(2):87-99. doi: 10.1002/pri.1599. Epub 2014 Jul 3. PMID 24996117
- [Background] Hektoen LF, Saltvedt I, Sletvold O, Helbostad JL, Luras H, Halsteinli V. One-year health and care costs after hip fracture for home-dwelling elderly patients in Norway: Results from the Trondheim Hip Fracture Trial. Scand J Public Health. 2016 Dec;44(8):791-798. doi: 10.1177/1403494816674162. Epub 2016 Oct 23. PMID 28929932
- [Result] Taraldsen K, Thingstad P, Dohl O, Follestad T, Helbostad JL, Lamb SE, Saltvedt I, Sletvold O, Halsteinli V. Short and long-term clinical effectiveness and cost-effectiveness of a late-phase community-based balance and gait exercise program following hip fracture. The EVA-Hip Randomised Controlled Trial. PLoS One. 2019 Nov 18;14(11):e0224971. doi: 10.1371/journal.pone.0224971. eCollection 2019. PMID 31738792